CLINICAL TRIAL: NCT05165082
Title: The Efficacy of Topical Timolol Combined With Cryotherapy in EGFR Inhibitor-induced Paronychia - a Double-blinded, Intrapatient Left-to-right Controlled Study
Brief Title: The Efficacy of Topical Timolol Combined With Cryotherapy in EGFR Inhibitors-induced Paronychia - a Double-blinded, Intrapatient Left-to-right Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Huang Yu Chen, Yu-Chen Huang, MD, Principal Investigator, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N202104033
Record Dates: First submitted 2021-11-10; First posted 2021-12-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Paronychia; Epidermal Growth Factor Receptor Inhibitor
MeSH Terms: conditions — Paronychia | interventions — Timolol; Ophthalmic Solutions; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Timolol plus cryotherapy (Experimental): Apply topical timolol solution twice daily (since the beginning of the allocation and continue for 8 weeks) and cryotherapy with liquid nitrogen once every other week (on the allocation day, at the 2nd week, 4th week and 6th week after the beginning of the trial).
  Interventions: Drug: Timolol maleate 0.5% ophthalmic solution; Procedure: Cryotherapy with liquid nitrogen
- Placebo plus cryotherapy (Placebo Comparator): Apply placebo (normal saline) twice daily (since the beginning of the allocation and continue for 8 weeks) and cryotherapy with liquid nitrogen once every other week (on the allocation day, at the 2nd week, 4th week and 6th week after the beginning of the trial).
  Interventions: Procedure: Cryotherapy with liquid nitrogen

INTERVENTIONS:
Drug: Timolol maleate 0.5% ophthalmic solution — Apply on affected finger or toes twice daily for 8 weeks
  Other Names: Timoptol
  Arms: Timolol plus cryotherapy
Procedure: Cryotherapy with liquid nitrogen — Conducted on affected finger or toes every other week for four sessions.

SUMMARY:
Background: EGFR inhibitors (EGFRi) have been used to treat a wide variety of cancers nowadays. One of the major side effects of EGFRi is paronychia, which was not fatal but may caused huge negative impact on patient's daily activities. Current guidelines regarding EGFRi-induced paronychia suggested treatment with cryotherapy, topical corticosteroid or surgical intervention for Common Terminology Criteria for Adverse Events (CTCAE) grade 2 to grade 3 lesions. Recent studies showed that topical beta-blockers may be effective treatment for EGFRi- induced paronychia. However, the evidence was limited to case series and there was no randomized trials evaluating the efficacy.

Goal: To evaluate whether topical timolol combined with cryotherapy was more effective than cryotherapy alone in treating EGFR inhibitors-induced paronychia.

Method: In this single center, randomized, double-blinded, left-to-right comparison study, we plan to enroll 35 patients with EGFR inhibitors-induced paronychia. Patients eligible to enter this study should be over the age of 20 having at least one finger or toe involved with CTCAE grade 2~3 paronychia on each of their hands or feet. The paronychia should have no indication for surgical treatment. After enrollment, one physician will randomize the hands or feet to either timolol-plus-cryotherapy group or cryotherapy-alone group using a computer-generated random allocation scheme. The side allocated to the timolol-plus-cryotherapy group will receive topical timolol solution twice daily (since the beginning of the allocation and continue for 8 weeks) and topical cryotherapy with liquid nitrogen every other week (at the allocation day, at the 2nd week, 4th week and 6th week after the beginning of the trial). The other side allocated to cryotherapy-alone group will receive placebo (normal saline) twice daily (since the beginning of the allocation and continue for 8 weeks) and topical cryotherapy with liquid nitrogen every other week (at the allocation day, at the 2nd week, 4th week and 6th week after the beginning of the trial). In the treatment phase, patients may receive additional local or systemic antibiotics according to the dermatologist's clinical judgement, but they can not receive topical silver nitrate, trichloroacetic acid or corticosteroid ointment. Patients are evaluated at baseline, at 2, 4, 6 and 8 weeks after the initiation of treatment. Efficacy endpoints include CTCAE grade, scoring system for paronychia related to oncologic treatments (SPOT) and physician global assessment, which are evaluated by a blinded investigator based on digital photos, and pain VAS score and patient global assessment, which are evaluated by questionnaire to the patients.

ELIGIBILITY:
Inclusion Criteria:

* EGFR inhibitors-induced paronychia
* Older than 20 years
* Having at least one finger or toe involved with CTCAE grade 2~3 paronychia on each of their hands or feet

Exclusion Criteria:

* Indication for surgical treatment
* Medical history of asthma, severe COPD, sinus bradycardia, SA block, 2nd to 3rd degree AV conduction delay, heart failure, cariogenic shock or allergy to timolol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at baseline
  The SPOT evaluates severity of each hand or foot based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. In each parameter, the finger (or toe) with the highest score was selected to be representative of the hand (or foot), and the sum of the four parameters makes the total score of the hand or foot. The highest score of each parameter could originate from different fingers (or toes). The total score of each hand (or foot) ranges from 0 to 12.
Scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at week 2 after the initiation of intervention
  The SPOT evaluates severity of each hand or foot based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. In each parameter, the finger (or toe) with the highest score was selected to be representative of the hand (or foot), and the sum of the four parameters makes the total score of the hand or foot. The highest score of each parameter could originate from different fingers (or toes). The total score of each hand (or foot) ranges from 0 to 12.
Scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at week 4 after the initiation of intervention
  The SPOT evaluates severity of each hand or foot based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. In each parameter, the finger (or toe) with the highest score was selected to be representative of the hand (or foot), and the sum of the four parameters makes the total score of the hand or foot. The highest score of each parameter could originate from different fingers (or toes). The total score of each hand (or foot) ranges from 0 to 12.
Scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at week 6 after the initiation of intervention
  The SPOT evaluates severity of each hand or foot based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. In each parameter, the finger (or toe) with the highest score was selected to be representative of the hand (or foot), and the sum of the four parameters makes the total score of the hand or foot. The highest score of each parameter could originate from different fingers (or toes). The total score of each hand (or foot) ranges from 0 to 12.
Scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at week 8 after the initiation of intervention
  The SPOT evaluates severity of each hand or foot based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. In each parameter, the finger (or toe) with the highest score was selected to be representative of the hand (or foot), and the sum of the four parameters makes the total score of the hand or foot. The highest score of each parameter could originate from different fingers (or toes). The total score of each hand (or foot) ranges from 0 to 12.

SECONDARY OUTCOMES:
Pain visual analogue scale | Evaluated at baseline, week 2, 4, 6 and 8 after the initiation of intervention
  Patients rate their severity of pain on a scale of 0 to 10, with 0 for no pain, 5 for moderate pain, and 10 for the worst pain ever experienced.
Physician global assessment | Evaluated at week 2, 4, 6 and 8 after the initiation of intervention
  The physician rates the improvement of lesions based on digital photographs on a scale of 0 to 6, representing:
  0, total clearance (100% improvement);
  1. almost total clearance (90% improvement);
  2. distinct clearance (75% improvement);
  3. moderate clearance (50% improvement);
  4. mild clearance (25% improvement);
  5. no change;
  6. worse.
Patient global assessment | Evaluated at week 2, 4, 6 and 8 after the initiation of intervention
  Patients rate their extent of improvement of lesions on a scale of 0 to 10, with 0 for no improvement, 5 for moderate improvement, and 10 for total clearance of lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Municipal Wan-Fang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu CY, Chen KY, Wen-Cheng Chang J, Wei YF, Lee CH, Wang WM. Taiwanese Dermatological Association consensus for the prevention and management of epidermal growth factor receptor tyrosine kinase inhibitor-related skin toxicities. J Formos Med Assoc. 2017 Jun;116(6):413-423. doi: 10.1016/j.jfma.2017.03.001. Epub 2017 Mar 27. PMID 28351555
- [Background] Yen CF, Hsu CK, Yang HS, Lee CN, Chi CC, Chung WH, Wang CL, Pang JS, Wang CW, Ko YS, Lu CW. Treatment of epidermal growth factor receptor inhibitor-induced severe paronychia with pyogenic granuloma-like lesions with topical betaxolol: an open-label observation study. Int J Dermatol. 2020 Mar;59(3):326-332. doi: 10.1111/ijd.14730. Epub 2019 Nov 25. PMID 31763692